CLINICAL TRIAL: NCT02237599
Title: A Feasibility Study of Integrated SSEP and Detection Algorithm for Detection of Intraoperative Positional Neuropraxia
Brief Title: Somatosensory Evoked Potential Algorithm for Detection of Intraoperative Positional Neuropraxia
Acronym: EPAD
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, John Murkin, PI, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 104826
Record Dates: First submitted 2014-07-17; First posted 2014-09-11 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Neuropraxia
Keywords: SSEP; neuropraxia; intraoperative; automated

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study hypothesizes that an automated device using small electronic impulses can detect nerve impairment in unconscious patients.

DETAILED DESCRIPTION:
Application of SSEP probes to bilateral ulnar and popliteal nerve areas with sensors at (1) bilateral brachial plexus (clavicles), (2) Erb's point (posterior C8 cervical spine) and (3) on forehead will permit microvolt current to to be detected and analyzed against a proprietary algorithm. Neuropraxia will be detected based on abnormalities developing in received SSEP signals.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery

Exclusion Criteria:

* neuromuscular disease stroke

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intraoperative adult patients undergoing surgical procedure
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2014-09; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Neuropraxia | postoperative
  Correlation between postoperative neuropraxia and intraoperative alert of impaired neural transmission detected via EPAD

CONTACTS AND LOCATIONS:
Overall Officials: John M Murkin, MD, Principal Investigator — Western University
Locations (1):
- University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No